CLINICAL TRIAL: NCT05504993
Title: Are Comorbidities Related to Frequent Severe Exacerbations of AECOPD
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Deniz Doğan Mülazimoğlu, University Lecturer, Ankara University
Other Study IDs: 05-305-18
Record Dates: First submitted 2022-08-14; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Chronic Obstructive Lung Disease; Acute Exacerbation of COPD; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High comorbidity group: CCI equal or higher than 2 COTE equal or higher than 4 COMCOLD equal or higher than 4
  Interventions: Other: Frequency of AECOPD
- Low comorbidity group: CCI lower than 2 COTE lower than 4 COMCOLD lower than 4
  Interventions: Other: Frequency of AECOPD

INTERVENTIONS:
Other: Frequency of AECOPD — No intervention has been applied. 92 COPD patients divided into 2 groups according to their comorbidity level. Than these groups were compared for their AECOPD frequency

SUMMARY:
INTRODUCTION: Relationship between comorbidities and COPD is two-sided. While the number of comorbidities increasing, the frequency of acute exacerbations of COPD (AECOPD) is increasing, too. Comorbidity indexes can be used for recognition of comorbidities while managing COPD patients. In the present study, it is aimed to compare comorbidity indexes such as Charlson Comorbidity Index, COMCOLD and COTE in the matter of exacerbation frequency.

METHOD: Subjects hospitalized for AECOPD, admitted to the study. Exacerbation severity, frequency, further exacerbations for a 1-year period in the follow-up period and CCI, COMCOLD and COTE scores were recorded. High and low comorbidity groups were compared for AECOPD frequency, severity, and further exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Admitted to the ward for AECOPD

Exclusion Criteria:

* Not giving informed consent
* Unable to perform PFT
* Lost to follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study included all patients, admitted to pulmonary diseases department, and hospitalized in ward for acute exacerbation of COPD (AECOPD) for a six-month period.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Frequency of AECOPD | 1 year
  Frequency of AECOPD in the last one year

SECONDARY OUTCOMES:
Having at least one severe AECOPD | 1 year
  having at least one severe AECOPD in the last year
Frequency of AECOPD for the next one year | 1 year
  the number of AECOPD for 1 year period from the preceding admission, regardless of severity

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided